CLINICAL TRIAL: NCT03857334
Title: Plantar Fasciitis Treatment: Double Blinded Randomized Control Study of the Efficacy of an Injection of Platelet Rich Plasma (PRP) Versus an Infiltration of Corticosteroids
Brief Title: Efficacy of Platelet Rich Plasma in Plantar Fasciitis
Acronym: APOPLANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UF 8737
Record Dates: First submitted 2018-04-27; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Biological: Injection of autologous platelet rich plasma
- Arm B (Active Comparator)
  Interventions: Drug: Injection of cortivazol : Altim®

INTERVENTIONS:
Biological: Injection of autologous platelet rich plasma
  Arms: Arm A
Drug: Injection of cortivazol : Altim® — Corticosteroids
  Arms: Arm B

SUMMARY:
Plantar fasciitis is a common pathology among podiatry moreover the healing time takes several months.

The main aim of this study is to evaluate the efficacy of a injection of Platelet-Rich Plasma (PRP) versus corticosteroid injection.

ELIGIBILITY:
Inclusion Criteria:

* Plantar fasciitis
* Average VAS greater than or equal to 5/10
* Resistance of medical reference treatment

Exclusion Criteria:

* Other plantar lesion find on RMI
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mean daily pain measured with a visual analog scale from 0 to 10 | 6 months
  Comparison of pain intensity, measured with a visual analog scale from 0 to 10

SECONDARY OUTCOMES:
Pain intensity during the first steps of the day measured with a visual analog scale from 0 to 10 | 6 months
  Measured with a visual analog scale from 0 to 10
Pain intensity on direct compression measured with a visual analog scale from 0 to 10 | 6 months
  Constant intensity of the compression, measured with a visual analog scale from 0 to 10
Impairment of walking function | 6 months
  Foot function index

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hosîtal, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breton A, Leplat C, Picot MC, Aouinti S, Taourel P, Laffont I, Julia M, Cyteval C. Prediction of clinical response to corticosteroid or platelet-rich plasma injection in plantar fasciitis with MRI: A prospective, randomized, double-blinded study. Diagn Interv Imaging. 2022 Apr;103(4):217-224. doi: 10.1016/j.diii.2021.10.008. Epub 2021 Nov 26. PMID 34844893